CLINICAL TRIAL: NCT00230217
Title: Evaluation of Single Agent Rasburicase in Treatment/Prevention of Hyperuricemia Associated With Tumor Lysis Syndrome in Adult and Pediatric Patients With Lymphoma/Leukemia/Solid Tumor Malignancies at Their First Relapse or Refractory Disease
Brief Title: Study of Rasburicase as Treatment or Prevention of Hyperuricemia Associated With Tumor Lysis Syndrome in Patients With Relapsed or Refractory Lymphoma, Leukemia, or Solid Tumor Malignancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EFC5339; NCT00086918 (obsolete NCT alias); NCT00247767 (obsolete NCT alias)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Tumors; Hyperuricemia; Tumor Lysis Syndrome
Keywords: Relapse; Refracturing; Leukemia; Lymphoma; Solid Tumor
MeSH Terms: conditions — Neoplasms; Hyperuricemia; Tumor Lysis Syndrome; Recurrence; Leukemia; Lymphoma | interventions — rasburicase; Urate Oxidase

INTERVENTIONS:
Drug: Rasburicase (SR29142)

SUMMARY:
This is an open-label, multi-center study with 2 arms. The primary objective is to assess the response to treatment with rasburicase in 2 populations of adult and pediatric patients with lymphoma/leukemia/solid tumor malignancies, those previously treated with a uricolytic agent, and those not previously treated with a uricolytic agent at their first relapse or refractory disease.

DETAILED DESCRIPTION:
This is a multi-center, 2 arm, open-label study;

* Arm A: Patients previously treated with a uricolytic agent;
* Arm B: Patients not previously treated with a uricolytic agent.

Patients receive rasburicase for 5 days and begin chemotherapy 4-24 hours after the first dose of rasburicase. Patients are followed at 14 and 35 days, at 3 and 6 months and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Meets one of the following risk criteria for tumor lysis syndrome (TLS):

   A patient is at high risk for TLS if he/she presents with:
   * Hyperuricemia of malignancy (plasma uric acid > 7.5 mg/dL);
   * A diagnosis of a very aggressive lymphoma/leukemia based on the Revised European-American Lymphoma (REAL) classification of lymphoma/leukemia;
   * Acute myeloid leukemia (AML);
   * Chronic myeloid leukemia (CML) in blast crisis; or
   * High grade myelodysplastic syndrome (refractory anemia with excess blast, refractory anemia with excess blast in transformation, or chronic myelomonocytic leukemia) only if they have > 10% bone marrow blast and are given aggressive treatment similar to AML

   A patient is at potential risk for TLS if he/she presents with:
   * A diagnosis of an aggressive lymphoma/leukemia based on the REAL classification of lymphoma/leukemia plus 1 or more of the following criteria:

     * Lactate dehydrogenase (LDH) > 2 x upper limit of normal (ULN)(IU/L)
     * Stage III-IV disease
     * Stage I-II disease with 1 lymph node/tumor > 5 cm in diameter
2. Patients previously treated with a uricolytic agent or not at their first relapse or refractory disease
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-3. ECOG equivalent derived from Karnofsky performance scale 100-30 or Lansky performance score 100-30 (patients < or = 16 years of age) may also be used.
4. Life expectancy >3 months
5. Negative pregnancy test (females of child bearing potential) and use of effective contraceptive method (both males and females). A pregnancy test may be performed on serum or urine human chorionic gonadotropin (HCG).
6. Signed written informed consent

Exclusion Criteria:

1. History of established diagnosis of asthma or severe life-threatening atopic allergy
2. Hypersensitivity to uricases or any of the excipients
3. Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency or history of hemolysis indicative of G6PD deficiency
4. Pregnant or lactating
5. Concomitant treatment with any investigational drug
6. Planned treatment with rituximab
7. Receipt of rituximab within the 12 month period prior to study entry
8. Unwilling or unable to comply with the requirements of the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2004-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Positive response based on plasma uric acid levels. | up to 48 hours after last administration.

SECONDARY OUTCOMES:
safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- United States (7):
  - Alta Bates Comprehensive Cancer Center, Berkley, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Florida Health Science Center at Jacksonville, Jacksonville, Florida
  - New York Medical College, Valhalla, New York
  - University of Oklahoma HSC, Oklahoma City, Oklahoma
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - Mary Babb Randolph Cancer Center, Morgantown, West Virginia